CLINICAL TRIAL: NCT01167465
Title: A Clinical Observation to Assess the Safety and Consumers' Satisfaction of Moussik vs Desitin Creamy Ointment in Prophylaxis of Diaper Rash. A Single Blind, Multicenter, Randomized, Cross-over Study
Brief Title: Determination of Safety and Consumers' Satisfaction of Moussik Versus Desitin Creamy Ointment in Diaper Rash Prophylaxis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Trima, Israel Pharmaceutical Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Diaper Rash
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Diaper Rash
Keywords: Diaper Dermatitis; Diaper Rash; Erythema
MeSH Terms: conditions — Diaper Rash; Erythema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Moussik Diaper Rash Mousse — To be used as instructed
Other: Desitin Creamy Ointment — To be used as instructed

SUMMARY:
The purpose of this clinical observation is to evaluate the safety and consumers' satisfaction of Moussik vs Desitin Creamy ointment as a diaper rash protection product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female infants aged between 3-18 months who are routine users of disposable diapers

Exclusion Criteria:

* Children with symptoms of systemic disease or skin lesions.
* Children diagnosed as having diaper dermatitis at baseline
* Known hypersensitivity to any of the components of the trial preparations.
* Children suffering from atopic diseases.
* Children who have participated during the last month in another clinical trial.

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Six point erythema skin grade | After two weeks
  0 - Normal skin
  + - Questionable erthema not covering entire area
  1. - Definite erythema
  2. - Erythema and induration
  3. - Vesiculation
  4. - Blister reaction

SECONDARY OUTCOMES:
Visual analogue scale (VAS) from 0 to 10 | After two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kobi Shiff, MD, Principal Investigator